CLINICAL TRIAL: NCT02755064
Title: Relationship Between Gastric Emptying and Glycemic Variability in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adil Bharucha (Other)
Responsible Party: Sponsor-Investigator, Adil Bharucha, Consultant, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-008620; UL1TR000135 (NIH)
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — erythromycin lactobionate; Sodium Chloride; Erythromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Erythromycin lactobionate IV 2 mg/kg (Experimental): During the second visit, erythromycin was given as an initial bolus of 0.5 mg/kg over 10 min immediately before the meal. The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Thereafter, an infusion of 1.5 mg/kg was given over the next 50 min with the same infusion pump.
  Interventions: Drug: Erythromycin lactobionate; Drug: [13C]-Spirulina
- Erythromycin lactobionate IV 3 mg/kg (Active Comparator): During the second visit, erythromycin was given as an initial bolus of 0.5 mg/kg over 10 min immediately before the meal. The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points.Thereafter, an infusion of 1.5 mg/kg was given over the next 50 min with the same infusion pump.
  Interventions: Drug: Erythromycin lactobionate; Drug: [13C]-Spirulina
- Placebo IV (Placebo Comparator): Saline was given as an initial bolus over 10 min immediately before the meal. The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points. Thereafter, an infusion of saline was given over the next 50 min with the same infusion pump.
  Interventions: Drug: Placebo IV; Drug: [13C]-Spirulina
- Erythromycin Ethylsuccinate Suspension (Experimental): In Phase 2 of the study, subjects randomized to this arm will receive Erythromycin Ethylsuccinate Suspension 250 mg tid orally for a total period of 7 days. The GEBT was performed approximately on day 7. The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points.
  Interventions: Drug: [13C]-Spirulina; Drug: Erythromycin Ethylsuccinate Suspension
- Placebo Suspension (Placebo Comparator): In Phase 2 of the study, subjects randomized to this arm will receive an oral placebo prepared to mimic the Erythromycin Ethylsuccinate Suspension for a total period of 7 days. The GEBT was performed approximately on day 7. The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points.
  Interventions: Drug: [13C]-Spirulina; Drug: Placebo Suspension

INTERVENTIONS:
Drug: Erythromycin lactobionate — In Phase 1 of the study, during the second visit, erythromycin was given as an initial bolus of 0.5 mg/kg over 10 min immediately before the meal. Thereafter, an infusion of 1.5 or 2.5 mg/kg was given over the next 50 min with the same infusion pump. The goal of testing 2 different doses was not to assess dose-related effects but to compare glycemic indices against a spectrum of gastric emptying rates.
  Other Names: Erythrocin™ Lactobionate-IV
  Arms: Erythromycin lactobionate IV 2 mg/kg; Erythromycin lactobionate IV 3 mg/kg
Drug: Placebo IV — In Phase 1 of the study, during the second visit, saline was given as an initial bolus over 10 min immediately before the meal. Thereafter, an infusion of saline was given over the next 50 min with the same infusion pump.
  Other Names: Saline
  Arms: Placebo IV
Drug: [13C]-Spirulina — The subject consumed the test meal containing 13C-Spirulina in no more than 10 minutes. Breath samples were collected at baseline obtained upon completion of the meal and at 15, 30, 45, 60, 90, 120, 150, 180, and 240 minute time points.
  Other Names: Carbon-13 Spirulina Breath Test; Gastric Emptying Breath Test (GEBT)
Drug: Erythromycin Ethylsuccinate Suspension — In Phase 2 of the study, subjects randomized to this arm will receive Erythromycin Ethylsuccinate Suspension 250 mg tid orally for a total period of 7 days.
  Other Names: E.E.S.
  Arms: Erythromycin Ethylsuccinate Suspension
Drug: Placebo Suspension — In Phase 2 of the study, subjects randomized to this arm will receive an oral placebo prepared to mimic the Erythromycin Ethylsuccinate Suspension for a total period of 7 days.
  Arms: Placebo Suspension

SUMMARY:
With this study, the investigators hoped to learn if the rate at which food empties from the stomach affects blood sugar values. Using data from this study, we hope to improve our ability to control blood sugars in individuals with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
The study comprised 3 outpatient visits over a period of 11 days. Safety lab test were performed at the screening visit. At each visit, GE was evaluated by 13C-spirulina breath tests.

Phase 1:

After the baseline assessment (GE1), the second and third GE tests were performed during treatment with intravenous (GE2) and oral erythromycin (GE3) or placebo. Subject arrived fasting at each study visit. Prior to gastric emptying study, there was placement of an intravenous line. Subject continued to take insulin and other medications as usual. Subjects were required to do finger-stick glucose readings 4 times a day or as instructed by their physician. Subjects were provided with a log sheet to keep track of meal times, insulin dosing and times, glucose readings, and activities. Continuous glucose monitoring (CGM) and gastric emptying were evaluated for the duration of the study (11 days) and thrice respectively. GE was evaluated at baseline (GE1) and after randomized to intravenous saline, erythromycin (2 mg/kg) or erythromycin (3 mg/kg).

Phase 2:

Thereafter, patients were randomized to erythromycin ethyl succinate suspension (250 mg tid) or placebo for a total period of 7 days. GE3 was preferably performed on day 7, after oral erythromycin or placebo was started.

An EKG was performed at baseline to identify (and exclude) patients who have contraindications to erythromycin. An EKG was also repeated at the end of the study, i.e., on GE3 for safety. No change to insulin (apart from those that patients do with their self management skills) or other medications was made during this research study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant non-breastfeeding female volunteers with type 1 diabetes mellitus (T1 DM) undergoing a clinically-indicated continuous glucose monitoring (CGM) study (Women of childbearing potential may be enrolled if they use contraceptives throughout the length of the study).
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
* Glycated hemoglobin (A1c) < 8.5 %

Exclusion Criteria:

* Severe nausea or vomiting precluding study assessments
* Use of medications that alter GI motility e.g., narcotics, medications with significant anticholinergic effects, CYP-450 3A4 inhibitors, antibiotics (other than the experimental drug erythromycin), pramlintide or GLP-1 based therapy. Subjects using metoclopramide or erythromycin will be enrolled but these medications will be held for 7 days before CGM1 and GE1
* Pancreas transplantation
* Contraindications to erythromycin: i.e., 1) concomitant therapy with astemizole, cisapride, pimozide, or terfenadine; 2) hypersensitivity to erythromycin or any component of the product; Corrected QT interval on EKG >460 msec
* Known family history of sudden death or congenital QT prolongation
* Serum potassium and magnesium levels outside of normal range at screening or visit 1
* Patients with moderate or severe renal insufficiency, i.e., subjects with an eGFR < 60 mL/min/1.73 m^2)
* Patients who are allergic to eggs, wheat or milk or unwilling to consume these products.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Relationship between gastric emptying and glycemia | 11 days
  GE was measured by 13C spirulina GEBT. Glycemia was measured with continuous glucose monitoring.

SECONDARY OUTCOMES:
Number of subjects with delayed gastric emptying | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parthasarathy G, Kudva YC, Low PA, Camilleri M, Basu A, Bharucha AE. Relationship Between Gastric Emptying and Diurnal Glycemic Control in Type 1 Diabetes Mellitus: A Randomized Trial. J Clin Endocrinol Metab. 2017 Feb 1;102(2):398-406. doi: 10.1210/jc.2016-2809. PMID 27880079